CLINICAL TRIAL: NCT06402188
Title: European ColoSeal™ ICD System Safety and Feasibility Study
Brief Title: ColoSeal™ ICD System Safety and Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Averto Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN0001
Record Dates: First submitted 2023-05-07; First posted 2024-05-07 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
Keywords: Colon anastomosis; Rectosigmoid cancer resection; Ostomy; Colon diversion
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- ColoSeal ICD Device Treatment Arm (Experimental): Subjects will undergo transanal placement of the ICD Device.
  Interventions: Device: ColoSeal ICD Device

INTERVENTIONS:
Device: ColoSeal ICD Device — The subject will undergo scheduled resection per the surgeon's preferred technique. Following completion of the anastomosis, the Intraluminal Colonic Diversion (ICD) Device will be inserted, advanced and positioned with the ICD Delivery System transanally. The ICD Device will remain in place for 10± 2 days. Anastomotic leak testing will be performed prior to scheduled removal.

SUMMARY:
The purpose of this clinical investigation is to evaluate the safety and feasibility of the ColoSeal ICD System in a prospective, multicenter, single-arm study. The ColoSeal ICD System is intended to be used to protect a damaged segment of colon such as a surgical anastomosis, anastomosis leak, or perforation from contact with fecal flow for up to 21 days. The device will be evaluated in adult patients with rectal and rectosigmoid cancer undergoing a resection with a colorectal anastomosis.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to evaluate the safety and feasibility of the ColoSeal ICD System in a prospective, multicenter, single-arm study. The ColoSeal ICD System is intended to be used to protect a damaged segment of colon such as a surgical anastomosis, anastomosis leak, or perforation from contact with fecal flow for up to 21 days. The device will be evaluated in adult patients with rectal and rectosigmoid cancer undergoing a resection with a colorectal anastomosis. Subjects will undergo scheduled resection per the surgeon's preferred technique. Following completion of the colon anastomosis, a leak check will be performed prior to insertion of the ColoSeal ICD Device to confirm no leak is present. The ICD Device will be inserted, advanced and positioned with the ICD Delivery System transanally. The anchor portion is positioned > 5 cm above and ideally 10-20 cm above (more proximal in GI tract) the area requiring protection from fecal flow (the anastomosis). The anchor portion of the device is designed to be placed in healthy bowel and not at the region of damaged bowel where protection is required. After positioning, deployment, and anchoring of the ICD Device the Delivery System is removed. The external portion of the device is further anchored to the subject's skin using an adhesive dressing and an optional extension tubing. The ICD Device will remain in place for 10+/-2 days post-operatively. An anastomosis leak test will be performed prior to device removal. Once no leak is confirmed, the ICD Device will be removed from the subject.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-65 years of age at screening, or subject is 66-70 years of age at screening with up to one cardiovascular, metabolic or pulmonary comorbidity for which medication is prescribed.
* Subject is diagnosed with rectosigmoid or rectal cancer
* Subject is scheduled for elective resection, either open, laparoscopic or robotic with mesorectal excision (either abdominal or transanal approach) which will require the creation of an anastomosis and protective ostomy (anastomosis maximally 15 cm from the anal verge).
* The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the appropriate Medical Ethics Committee (EC) or Institutional Review Board (IRB).
* Subject must be willing and able to comply with study follow-up requirements.

Exclusion Criteria:

* Subject with a life expectancy < 1 year
* Subjects with ASA classification > 3
* Albumin < 30 g/liter
* Subject has local or systemic infection at the time of intervention.
* Major surgical or interventional procedures within 30 days prior to this study or planned major surgical or interventional procedures within 1 month of entry into this study
* Patient has received systemic chemotherapy or radiation to the pelvis within 30 days prior to the planned procedure
* Subject has a diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, ischemic bowel, carcinomatosis, diverticulitis, or extensively spread inflammatory bowel disease
* Subjects has a diagnosis of coagulopathy, thrombocytopenia, immune suppression
* BMI ≥ 40
* Subject is scheduled for a concurrent major surgical procedure during the surgery (e.g., liver resection)
* Subject has been taking regular systemic/ steroid medication in the last 3 months
* Subjects is taking antimetabolites or antiplatelet agents
* Subject has undergone a prior pelvic anastomosis
* Subject requires an end-to-end anastomosis smaller than 31 mm in diameter
* Known allergy to any component of the device
* Known allergy to iodine or iodine-based contrast
* Any condition or abnormality which in the opinion of the investigator may jeopardize the subject's safe participation or the quality of the data
* Subject is pregnant or planning to become pregnant. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to surgical procedure
* Subject is unable or unwilling to provide informed consent
* Subject is currently participating in an investigational drug or another device study that clinically interferes with the current study endpoints

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with device related adverse events | 90 days post procedure
  Any device related adverse events during procedure and/or follow-up

SECONDARY OUTCOMES:
Procedure success | Day 0
  Rate of acute efficacy in placing and deploying the device at the desired location
Procedure time | Day 0
  Time from insertion of the introducer to the vacuum system being ready to be connected and begin vacuum application
Migration rate | Up to 21 days
  Number of devices migrated over the anastomosis divided by the number of devices placed
Occurrence of anastomotic leakage | Up to 90 days post procedure
  Anastomotic leak rate will be defined as any anastomotic leak during study follow-up period identified on radiographic analysis. Clinically symptomatic and non-symptomatic leaks (radiographically diagnosed only) will be analyzed separately and taken into account during comparative analysis to rates reported in literature. Anastomotic leak rate will be subdivided into those leaks occurring while device is in place in subject or late leaks after device removal.
Need for ostomy surgery | Up to 90 days post procedure
  Efficacy will be determined by ostomy avoidance rate. Need for ostomy percentage will be defined as the total number of subjects that required ostomy during study follow-up period over total number of subjects enrolled who would have a planned ostomy if not a study participant.
Successful device removal | Up to 21 days
  Percent of successful device removals without adverse effect

CONTACTS AND LOCATIONS:
Overall Officials: Hurshid Djamshidovich, MD, Principal Investigator — National Cancer Institute Tashkent Uzbekistan
Locations (3):
- National Center of Oncology after V.A. Fanarjian, Yerevan, Armenia
- Israeli-Georgian Medical Research Clinic Healthycore, Tbilisi, Georgia
- National Cancer Institute, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No